CLINICAL TRIAL: NCT00005959
Title: Phase II Trial of Rituximab in Combination With CHOP Chemotherapy in Patients With Previously Untreated Intermediate or High Grade Non-Hodgkin's Lymphoma
Brief Title: Combination Chemotherapy Plus Rituximab in Treating Patients With Intermediate-Grade or High-Grade Non-Hodgkin's Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Amgen (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067940; AMGEN-GCSF-990756; NCI-V00-1593
Record Dates: First submitted 2000-07-05; First posted 2003-12-17 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2002-06

CONDITIONS: Lymphoma
Keywords: stage III grade 3 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult Burkitt lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult Burkitt lymphoma; contiguous stage II grade 3 follicular lymphoma; contiguous stage II adult diffuse small cleaved cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; contiguous stage II adult diffuse large cell lymphoma; contiguous stage II adult Burkitt lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult Burkitt lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma | interventions — Filgrastim; Rituximab; Cyclophosphamide; Doxorubicin; Prednisone; Vincristine

INTERVENTIONS:
Biological: filgrastim
Biological: rituximab
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: prednisone
Drug: vincristine sulfate

SUMMARY:
RATIONALE: Monoclonal antibodies such as rituximab can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one chemotherapy drug with rituximab may kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of rituximab plus combination chemotherapy in treating patients who have intermediate-grade or high-grade non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the rate of complete response and partial response in patients with intermediate or high grade non-Hodgkin's lymphoma treated with rituximab plus cyclophosphamide, doxorubicin, vincristine, and prednisone (CHOP). II. Determine the toxicity of this regimen in these patients. III. Determine the disease-free and overall survival, time to response, and time to disease progression in patients treated with this regimen.

OUTLINE: This is a multicenter study. Patients are stratified according to the number of risk factors (0-2 vs 3-5). Risk factors include age (no greater than 60 vs greater than 60), tumor stage (II vs III or IV), number of extranodal sites (no more than 1 vs more than 1), performance status (0-1 vs 2-4), and serum LDH level (no greater than normal vs greater than normal). Patients receive rituximab IV on day 1; cyclophosphamide, doxorubicin, and vincristine IV on day 3; and oral prednisone on days 3-7. Patients over 60 also receive filgrastim (G-CSF) subcutaneously beginning on day 4 and continuing until blood counts recover (all other patients receive G-CSF as secondary prophylaxis). Treatment continues every 3 weeks for 4 courses in the absence of disease progression or unacceptable toxicity. Patients who respond receive 2 more courses. Patients who have no measurable disease after 6 courses receive rituximab IV once weekly for 4 consecutive weeks. This treatment continues every 6 months for 4 courses in the absence of disease progression or unacceptable toxicity. Patients who have measurable disease after 6 courses of chemotherapy receive 2 more courses for a maximum of 8 courses of CHOP, followed by maintenance therapy with rituximab (as described above). Patients are followed every 6 months for 2 years.

PROJECTED ACCRUAL: Approximately 100 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed intermediate or high grade non-Hodgkin's lymphoma Stage II, III, or IV disease B-cell where lymphoid cells are CD20 or CD19 positive No mantle cell, lymphoblastic, or peripheral T-cell non-Hodgkin's lymphoma Measurable or evaluable disease No prior treatment for lymphoma No known CNS metastases A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 60-100% Life expectancy: At least 12 weeks Hematopoietic: Unless documented bone marrow disease: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: SGOT and SGPT no greater than 3 times upper limit of normal Bilirubin no greater than 1.5 mg/dL Renal: Creatinine no greater than 2.0 mg/dL Cardiovascular: No history of severe heart disease, cardiomyopathy, or congestive heart failure LVEF normal by MUGA or echocardiogram Other: Not pregnant or nursing Fertile patients must use effective contraception No active infection as defined by: Clinical syndrome consistent with a viral or bacterial infection (e.g., influenza, upper respiratory infection, urinary tract infection) OR Fever with a clinical site of infection identified OR Microbiologically documented infection, including, but not limited to, bacteremia or septicemia No known HIV positivity No known sensitivity to E. coli derivatives (e.g., asparaginase, human insulin, human growth hormone, interferon alfa-2b) No other prior malignancy within the past 5 years except surgically cured basal or squamous cell skin cancer or carcinoma in situ of the cervix No psychiatric, addictive, or other disorder that may preclude study

PRIOR CONCURRENT THERAPY: Biologic therapy: See Disease Characteristics No concurrent biologic therapy except epoetin alfa No white blood cell transfusions Chemotherapy: See Disease Characteristics No concurrent chemotherapy Endocrine therapy: Not specified Radiotherapy: See Disease Characteristics No concurrent radiotherapy Surgery: At least 2 weeks since prior major surgery Other: No other concurrent investigational therapy No prophylactic antibiotics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-12

CONTACTS AND LOCATIONS:
Overall Officials: Carol Brannan, BS, BSN, Study Chair — Amgen
Locations (27):
- United States (27):
  - Montgomery Cancer Center, Montgomery, Alabama
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Providence Saint Joseph Medical Center - Burbank, Burbank, California
  - Cancer and Blood Institute of the Desert, Rancho Mirage, California
  - Southeast Florida Hematology-Oncology Group, Fort Lauderdale, Florida
  - Oncology-Hematology Group of South Florida, Miami, Florida
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - Hematology-Oncology Associates, PA, Pensacola, Florida
  - Hutchinson Clinic, P.A., Hutchinson, Kansas
  - Hematology/Oncology Care Inc., Crestview Hills, Kentucky
  - Maine Center for Cancer Medicine and Blood Disorders, Scarborough, Maine
  - Associates in Oncology and Hematology, Rockville, Maryland
  - North Shore Cancer Center, Peabody, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Lakeland Medical Center - St. Joseph, Saint Joseph, Michigan
  - Bond Clinic, Rolla, Missouri
  - Midwest Hematology Oncology Consultants, Ltd., St Louis, Missouri
  - Hematology Oncology Associates, Morristown, New Jersey
  - New Mexico Oncology-Hematology, Albuquerque, New Mexico
  - HemOnCare, P.C., Brooklyn, New York
  - Our Lady of Mercy Medical Center, The Bronx, New York
  - N.W. Carolina Oncology & Hematology, P.A., Hickory, North Carolina
  - Oncology/Hematology Care, Inc., Cincinnati, Ohio
  - University of Tennessee, Memphis, Memphis, Tennessee
  - Intermountain Hematology/Oncology Associates, Inc., Salt Lake City, Utah
  - Vermont Center for Cancer Medicine, Inc., Colchester, Vermont
  - Hematology & Oncology Associates of Virginia, Richmond, Virginia